CLINICAL TRIAL: NCT04945005
Title: Prevention of Pacemaker Lead Induced Tricuspid regurgitAtion by Transesophageal eCho guidEd Implantation Registry
Acronym: PLACE
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Daniel Braun, MD, Attending Physician, LMU Klinikum
Other Study IDs: 101214
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Tricuspid Valve Insufficiency; Pacemaker Complication; Echocardiography, Transesophageal
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lead implantation with transesophageal echocardiography: All patients undergoing pacemaker/CRT implantation with concomitant transesophageal echocardiography in addition to fluoroscopic guidance
  Interventions: Procedure: Transesophageal guidance of lead implantation
- Lead implantation without transesophageal echocardiography (retrospective): All patients undergoing standard pacemaker/CRT implantation guided by fluoroscopy only (retrospective historical control group)

INTERVENTIONS:
Procedure: Transesophageal guidance of lead implantation — In patients undergoing lead implantation including transesophageal echocardiography for clinical reasons (e.g. intraprocedural cardioversion), echocardiography was also used for guidance of lead implantation to reduce lead-leaflet interactions
  Groups: Lead implantation with transesophageal echocardiography

SUMMARY:
Registry for patients undergoing pacemaker/ICD implantation including a transtricuspid lead with and without intraprocedural transesophageal echocardiography to evaluate risk factors for lead induced tricuspid regurgitation.

DETAILED DESCRIPTION:
Lead induced tricuspid regurgitation is a common finding after pacemaker/ICD Implantation. Transesophageal echocardiography (TEE) might be used to guide lead implantations in order to prevent tricuspid regurgitation.

In this registry, patients undergoing pacemaker/ICD implantation including a transtricuspid lead are enrolled. While in most patients lead implantation is guided by fluroscopy, in some patients lead implantation is guided by TEE in addition to fluroscopy.

Aims of this registry: Evaluation of

* Incidence of lead induced tricuspid regurgitation
* Mortality and morbidity of lead induced tricuspid regurgitation
* Identification of risk factors for lead induced tricuspid regurgitation
* Influence of the lead position within the tricuspid valve on the incidence of lead induced tricuspid regurgitation
* Prevention of lead induced tricuspid regurgitation by TEE-guided lead implantation

ELIGIBILITY:
Inclusion Criteria:

* indication for pacemaker/ICD implantation including a transtricuspid lead according to guidelines

Exclusion Criteria:

* pre-existing RV lead
* pre-existing TR >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing pacemaker/ICD implantation including a transtricuspid lead were included in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Increase of tricuspid regurgitation by at least one grade (on a scale from 0-4) | 2 - 7 days post-implant (at hospital discharge)
  Lead induced tricuspid regurgitation measured by transthoracic echocardiography

SECONDARY OUTCOMES:
Dose-are product | Intraprocedural
  Dose-are product applied during lead implantation
Lead revisions | 30 days
  Incidence of acute lead revisions within 30 days
Increase of tricuspid regurgitation by at least one grade (on a scale from 0-4) | 3 months
  Lead induced tricuspid regurgitation measured by transthoracic echocardiography
Increase of tricuspid regurgitation by at least one grade (on a scale from 0-4) | 12 months
  Lead induced tricuspid regurgitation measured by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Braun, PD Dr. med., Principal Investigator — LMU Klinikum
Locations (1):
- LMU Klinikum, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gmeiner J, Sadoni S, Orban M, Fichtner S, Estner H, Massberg S, Hagl C, Nabauer M, Hausleiter J, Braun D. Prevention of Pacemaker Lead-Induced Tricuspid Regurgitation by Transesophageal Echocardiography Guided Implantation. JACC Cardiovasc Interv. 2021 Dec 13;14(23):2636-2638. doi: 10.1016/j.jcin.2021.08.042. No abstract available. PMID 34887055